CLINICAL TRIAL: NCT06547905
Title: Evaluation of an Ostomy Leakage Detection System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6028-OST
Record Dates: First submitted 2024-06-14; First posted 2024-08-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leakage Detection System arm (Experimental): Participants will utilize the leakage detection system
  Interventions: Device: Ostomy Leakage Detection System

INTERVENTIONS:
Device: Ostomy Leakage Detection System — A system that is used to detect ostomy leaks

SUMMARY:
This study will evaluate the safety and efficacy of an ostomy leakage detection system.

DETAILED DESCRIPTION:
Individuals with an ostomy will be recruited to evaluate an ostomy leakage detection system. The ostomy leakage detection system is designed to detect leaks and notify users of the leaks. Participants will evaluate the safety and efficacy of the leakage detection system.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or Older
2. Currently resides in the United Kingdom
3. Has an ileostomy, colostomy, or urostomy
4. Has a stoma diameter within the following range: 15 mm - 70 mm
5. Has a mild or moderate peristomal skin complication as defined using the Ostomy Skin Tool (OST) 2.0 (decision tree (DT)=1 or DT=2).
6. Has experienced a leak underneath or outside the perimeter of the barrier in the last 30 days or has worried about leakage in the last 30 days
7. Willing to use their typical ostomy pouching system together with the study product for duration of study
8. Currently has an Android Smart phone or an Apple iPhone of the following operating systems (OS):

   * a. Android Devices:

     * i. Compatible Brands: Samsung Galaxy, Huawei, Google Pixel
     * ii. Operating System: Android OS 9.0 (Pie) and later
   * b. Apple iPhones:

     * i. Compatible Models: iPhone X and later
     * ii. Operating System: iPhone Operating System (iOS) 15 and newer
9. Is willing to download the phone application for use during the study
10. Is willing to follow protocol procedures, as indicated by signing the informed consent
11. Is able to receive, read, and respond to English surveys electronically (i.e. via a computer or smart phone)

Exclusion Criteria:

1. Subject reports changing their ostomy barrier 3 or more times per day in the last 30 days
2. Has an electrical implant (e.g. pacemaker or internal defibrillator) and/or body worn medical device (e.g. insulin pump)
3. Subject reports that a caregiver, or someone other than themselves, is solely responsible for changing their ostomy pouching system. Note: subjects that use a combination of self-care and other assistance should not be excluded.
4. Reports as legally blind and/or deaf
5. Subject does not report a peristomal skin complication (PSC) or the subject reports a PSC that is scored as severe on the OST 2.0 tool (either a DT=0 or DT=3).
6. Subject reports currently having an abdominal fistula or abdominal wound
7. Subject has more than one stoma
8. Is undergoing chemotherapy, radiation, or non-inhaled steroid therapy (topical/applied to the skin around the stoma) that may compromise the skin
9. Is pregnant or breastfeeding at time of eligibility, as determined by self-report. Note: this exclusion will not be re-confirmed throughout the study after eligibility.
10. Is currently involved in another research study involving use of ostomy study products or accessories
11. Is currently an employee of a Company that manufactures Ostomy Products and/or Ostomy Accessories

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
The Accuracy of the Leakage Detection System (LDS) | through study completion, approximately 1 month
  The frequency of true positive, true negative, false positive, and false negative leakage detection events will be used to quantify the accuracy of the leakage detection system.

SECONDARY OUTCOMES:
How adherent subjects are to leakage notifications (ratio) | through study completion, approximately 1 month
  The proportion of barriers that are changed due to accurate leakage notifications will yield insights into how adherent subjects are to leakage notifications.
How efficacious leakage detection and notification was at alerting subjects to catastrophic leaks (ratio) | through study completion, approximately 1 month
  The ratio of the number of times subjects were alerted to leakage prior to a CL occurring to the number of times a barrier change was associated with a Catastrophic leak
Whether and to what extent the LDS affected Quality of Life (QoL), measured using the Ostomy leak Impact (OLI) validated tool | through study completion, approximately 1 month
  QoL will be measured at baseline and after approximately 1 month to determine whether the LDS affected QoL and to what extent using the OLI which is scored on a scale of 0-100 with higher scores indicating better outcomes
Whether and to what extent the LDS affected Quality of Life (QoL), measured using the Ostomy Adjustment Inventory-23 (OA1-23) validated tool | through study completion, approximately 1 month
  QoL will be measured at baseline and after approximately 1 month to determine whether the LDS affected QoL and to what extent using the OAI-23 which is scored on a scale of 0-92 with higher scores indicating better outcomes
Whether and to what extent the LDS affected Quality of Life (QoL), measured using the Single-item Sleep Quality Scale (SQS) validated tool | through study completion, approximately 1 month
  QoL will be measured at baseline and after approximately 1 month to determine whether the LDS affected QoL and to what extent using the SQS which is scored on a scale of 0-10 with higher scores indicating better outcomes

OTHER OUTCOMES:
Whether and to what extent the LDS affected peristomal skin health, measured by the Ostomy Skin Tool 2.0 (OST 2.0) validated tool | starting at day 0, every 7 days, through day 28
  The Ostomy Skin Tool 2.0 (OST 2.0) validated tool will be used to evaluate and compare skin health before subjects use the LDS at the Day 0 Periodic assessment and every 7 days thereafter up to Day 28. The OST 2.0 is scored on a scale of 0-3 with higher scores indicating worse outcomes.
Whether and to what extent the LDS affected healthcare resource utilization (HRU) and cost-effectiveness | through study completion, approximately 1 month
  Ostomy accessory usage, unplanned ostomy-related healthcare visits to a provider (such as a nurse or doctor, for example), incidence of and severity of PSCs (which have been shown to be associated with increased HRU), and/or wear (use) time of the ostomy barrier will be measured at periodic timepoints in the study (days 0, 7, 14, 21, 28, and/or 30) to obtain healthcare resource utilization (or cost) data which will be aggregated (summed) to evaluate the effect the LDS has on HRU and cost-effectiveness.
To evaluate how satisfied users were with the alerts/notifications from the LDS | through study completion, approximately 1 month
  Satisfaction scores will be reported as the proportion of each response option on a 5-point scale, from very unsatisfied to very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hugill, Principal Investigator — Dansac
Locations (1):
- PPD Development, L.P.; Decentralized, Virtual Site; 11 Granta Park, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No